CLINICAL TRIAL: NCT04286178
Title: The Effects of Exercise, Creatine, and Coenzyme Q10 Supplementation on Muscle Function in Children With Myositis
Brief Title: Exercise, Creatine and Coenzyme Q10 for Childhood Myositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian Feldman, Division Head, Division of Rheumatology, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1000062314; HC6-24-c228771 (Other: Health Canada)
Record Dates: First submitted 2020-02-06; First posted 2020-02-26 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Myositis, Juvenile
MeSH Terms: conditions — Dermatomyositis | interventions — Creatine; ubiquinol; coenzyme Q10; Glucose; Gels; Exercise

STUDY DESIGN:
Intervention Model Description: This study will be a double-blinded, placebo-controlled, randomized, multiple baseline design (MBD) where each subject will be randomly allocated a start time for the active supplements
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): patients in this arm will be treated with creatine and coenzyme Q10 supplements
  Interventions: Dietary Supplement: creatine monohydrate; Dietary Supplement: ubiquinol; Behavioral: Exercise
- Placebo (Placebo Comparator): patients in this arm will be given placebo supplements that look and taste identical to the active supplements
  Interventions: Dietary Supplement: glucose tablet; Dietary Supplement: gel capsule; Behavioral: Exercise

INTERVENTIONS:
Dietary Supplement: creatine monohydrate — Creatine will be taken at a dose of 150mg/kg/day of creatine base divided into 2 daily doses up to 39.7kg in body weight, after which dosing will be based on body surface area (BSA) at 4.69g/m2/day. Creatine will be administered orally as a chewable tablet provided by BioTechUSA™. Tablets are 2g and contain 0.9g of creatine monohydrate which is equivalent to 0.8g of creatine base.
  Arms: Treatment
Dietary Supplement: ubiquinol — Coenzyme Q10 (CoQ10, ubiquinol) will be taken at a dose of 10mg/kg/day divided into 2 daily doses with a daily maximum of 500mg. CoQ10 will be administered orally in 50mg softgels containing 50mg of ubiquinol (Active Q®), provided by Tishcon Corporation.
  Other Names: coenzyme Q10
  Arms: Treatment
Dietary Supplement: glucose tablet — Creatine placebo will be in the form of a glucose tablet with identical appearance and taste to the active supplement. The number of tablets/day will be determined based on the dose of creatine required for each patient.
  Arms: Placebo
Dietary Supplement: gel capsule — Ubiquinol placebo will be in the form of a gel capsule with identical appearance to the active supplement. The number of capsules/day will be determined based on the dose of ubiquinol required for each patient.
  Arms: Placebo
Behavioral: Exercise — Participants will be coached to hit 12,000 steps or 60 "active minutes" per day as logged by a FitBit (FitBit calculates active minutes as activities equivalent to moderate-to-vigorous physical activity (MVPA) done continuously for at least 10 minutes)

SUMMARY:
Children with JDM are weak and get tired because their muscles aren't able to work like healthy muscles. This can make it hard for them to do normal everyday things and can make them less happy about their lives compared to children without the disease. There are two nutritional supplements that help muscles use energy and recover after exercise: creatine and coenzyme Q10. If the muscle has more energy, it may not be as weak and may not feel as tired or sore after exercise. Because of this we want to see if having children with JDM take creatine and coenzyme Q10 can make them stronger and less tired. If this works, we hope it will let them be able to do the things that healthy children can do, and make them feel better about their lives.

ELIGIBILITY:
Inclusion Criteria:

* Ages 7 to 18 years
* Diagnosis of juvenile idiopathic inflammatory myopathy (JIIM) according to the 2017 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) criteria: ≥90% probability, age of onset <18 years
* Subjects on a stable course of medication (unlikely to change over study treatment period as determined by treating physician)
* Minimum height of 132.5cm (required to fit on the cycle ergometer)

Exclusion Criteria:

* Subjects with newly diagnosed JIIM within the previous 6 months
* Subjects unable to cooperate with study procedures, or too weak to participate in the exercise testing
* Subjects with impaired kidney function as determined from pre-baseline visit screening lab values (eGFR <90 ml/min/1.73m^2)
* Subjects currently taking anti-hypertensive drugs or blood thinners
* Subjects who are currently pregnant or planning to become pregnant within the study period

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Change in muscle function | 6 months
  Change in muscle function will be determined by the change in peak power achieved on the wingate anaerobic cycling test between the active supplement phase and the placebo phase

SECONDARY OUTCOMES:
Change in muscle fatigue | 6 months
  Change in muscle fatigue will be determined by the change in the fatigue index during the wingate test. Fatigue index is a percentage, and is calculated as follows: [(Peak Power - End Power)/Peak Power] x100
Change in general fatigue | 6 months
  Change in fatigue will be determined by the change in the Pediatric Quality of Life - Fatigue Module scores (PedsQL-Fatigue). This measure is scored on a scale of 0-100 with 100 representing the least amount of fatigue.
Change in quality of life | 6 months
  Change in quality of life will be determined by the change in the Quality of My Life questionnaire scores. Quality of my Life consists of 3 visual analog scales each scored out of 10. Higher scores indicate better quality of life.
Change in physical function | 6 months
  Change in physical function will be determined by the change in the hand grip strength, measured using a hand dynamometer. Three attempts will be given per hand, and the maximum grip strength achieved (in kg displaced) will be recorded for each hand.
Change in physical function | 6 months
  Change in physical function will be determined by the change in the vertical jump achieved, measured in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Brian Feldman, MD, MSc, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No